# **COVER PAGE**

## **Informed Consent Form**

OFFICIAL TITLE: Neoadjuvant Chemoradiotherapy and Consolidation Chemotherapy for Rectal Cancer: A Randomized Controlled Trial

**BRIEF TITLE:** Neoadjuvant Chemoradiotherapy and Consolidation Chemotherapy for Rectal Cancer

UNIQUE PROTOCOL ID: NCCCRC DOCUMENT DATE: August 2022

### **Principal Investigator:**

Konstantinos Perivoliotis, MD Telephone: 00302413501000 Email: kperi19@gmail.com

### **Sub-Investigators:**

Ioannis Baloyiannis Ioannis Samaras Athanasios Kotsakis Georgios Kyrgias

### **Study Director**

George Tzovaras, Professor of General Surgery

Telephone: 00302413502804 Email: gtzovaras@hotmail.com

> Department of Surgery University Hospital of Larissa Mezourlo 41110 Larissa Greece

# UNIVERSITY OF THESSALY, DEPARTMENT OF

UNIVERSITY GENERAL HOSPITAL OF LARISSA Mezourlo, 41110, Larissa

SURGERY CLINIC

**Director: Professor Zacharoulis Dimitrios** A 'Building, 2nd Floor, P.G.N. Of Larissa



### UNIVERSITY OF THESSALY, FACULTY OF MEDICINE

UNIVERSITY HOSPITAL OF LARISSA Mezourlo, 41110, Larissa GREECE

#### GENERAL SURGERY DPT

Chairman: Prof. Zacharoulis Dimitrios A 'Wing, 2nd Floor, University Hospital of Larissa

### **Research Protocol**:

# Neoadjuvant Chemoradiotherapy and Consolidation Chemotherapy for Rectal Cancer: A Randomized Controlled Trial

The purpose of this research protocol is to compare neoadjuvant chemoradiotherapy and consolidation chemotherapy with neoadjuvant chemoradiotherapy and adjuvant chemotherapy for rectal cancer. The study protocol is designed as a prospective randomized controlled study. The comparison of the two groups will be based on early and late postoperative endpoints. In addition, the efficacy of both approaches in terms of the specimen quality characteristics and the oncological outcomes will be evaluated.

### 1. Procedure

The patient will be admitted to the surgical department according to the predetermined procedure. All the necessary preoperative and laboratory examinations will be performed. A multidisciplinary oncology board will follow to determine the optimal treatment. The patient, then, will be randomized to one of the two groups. Following this, the patient will be submitted to the optimal operation for him / her to treat his / her condition. Postoperatively the patient will be monitored in the surgical department according to the existing protocols and guidelines.

### 2. Dangers

The risks are related to the possible postoperative complications from the operation.

### 3. Expected benefits

The research will result to the publication of data - results. Your participation in the protocol implies that you agree with future publication of results, provided that the information will be anonymous, and the names of the participants will not be disclosed. The data that will be collected will be encoded with a number, so that your name will not appear anywhere.

### 4. Information

Do not hesitate to ask questions regarding the purpose or the process of the protocol. If you have any doubts or questions, please ask us to give you clarifications.

### 5. Participation

Your participation in the protocol is voluntary. You are free to disagree or cancel your participation whenever you wish.

## 6. Informed consent

I have read this form and I understand the processes that I will follow. I agree to participate in the research protocol.

| Date:// |
|--------------------------------|
| Participant Name and Signature |

**Investigator Signature** 

**Principal Investigator:** Konstantinos Perivoliotis, MD

Telephone: 00302413501000 Email: kperi19@gmail.com

### **Study Director:**

George Tzovaras, Professor of General Surgery Telephone: 00302413502804 Email: gtzovaras@hotmail.com